CLINICAL TRIAL: NCT03117335
Title: Recombinant Endostatin With Vinorelbine and Cisplatin (NP) Plus Maintenance Therapy With Recombinant Endostatin for Advanced Non-small Cell Lung Cancer: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Study
Brief Title: Recombinant Endostatin Combined With Vinorelbine and Cisplatin in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Wuzhong Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG1107RHE; BA2010071 (Other Grant/Funding Number: Science and Technology Department of Jiangsu Province)
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Sulijia; Recombinant endostatin; Vinorelbine; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sodium Chloride; Endostatins

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vinorelbine plus Cisplatin With placebos (Active Comparator): The control group
  Interventions: Drug: Placebos
- Vinorelbine plus Cisplatin With Sulijia (Experimental): The treatment group
  Interventions: Drug: Sulijia

INTERVENTIONS:
Drug: Placebos — Drug 1:
  Placebo(Sodium Chloride Injection),7.5mg/m2 on d1-d14 in each 21-day cycle（stop interventing until the disease progress）
  Drug 2:
  Vinorelbine-Cisplatin:
  Vinorelbine, 25mg/m2, iv, on d1 and d8 in each 21-day cycle (no more than 4 cycles); Cisplatin,75mg/m2, iv, on d1 in each 21-day cycle(no more than 4 cycles)
  Other Names: Sodium Chloride Injection
  Arms: Vinorelbine plus Cisplatin With placebos
Drug: Sulijia — Drug 1:
  Sulijia(Recombinant Endostatin Injection) Sulijia, 7.5mg/m2 on d1-d14 in each 21-day cycle（stop interventing until the disease progress）
  Drug 2:
  Vinorelbine-Cisplatin:
  Vinorelbine, 25mg/m2, iv, on d1 and d8 in each 21-day cycle (no more than 4 cycles); Cisplatin,75mg/m2, iv, on d1 in each 21-day cycle(no more than 4 cycles)
  Other Names: Recombinant endostatin injection
  Arms: Vinorelbine plus Cisplatin With Sulijia

SUMMARY:
The main object of this trial is to offer treatment of recombinant endostatin ( Sulijia) combined with Vinorelbine and Cisplatin (NP) plus maintenance therapy with Sulijia for advanced Non-small Cell Lung Cancer, expecting to improve progression free survival (PFS) , disease control rate(DCR) , objective response rate(ORR) and Overall survival (OS) compared with chemotherapy alone, and evaluate the efficacy and safety of Sulijia.

DETAILED DESCRIPTION:
Recombinant endostatin injection Sulijia is a new type of recombinant protein drugs inhibiting tumor angiogenesis developed by a group of Chinese scientists and clinician. It is expressed in E. coli which Consists of 184 amino acids. It appears to be better than NP chemotherapy alone in terms of efficacy in phase I/II trials for advanced NSCLC. In this study, a randomized, double-blind, Placebo plus NP as control, multi-center phase III trial was designed to evaluate the safety and efficacy of Sulijia plus NP in the treatment of advanced NSCLC patients. PFS (progress free survival) is the primary end-point with OS (overall survival), ORR (objective response), DCR (disease control rate) and safety as the secondary end-point. A total of 560 patients have been recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 to 70 years old;
2. Patients with histological confirmed stage IV NSCLC;
3. According to the standard of RECIST1.1, they should have at least one of accurately measurable lesions with the largest diameter >=10mm by spiral CT, PET-CT, with the largest diameter >=20mm by ordinary CT and MRI;
4. general condition ECOG performance scale (PS) 0-1;
5. Life expectancy of more than 3 months;
6. No major organ dysfunction and laboratory indicators should meet the following requirements: absolute neutrophil count > 1.5*10^9/L, platelet count> 90*10^9/L, hemoglobin> 9g/dL; liver function: serum bilirubin was less than 2* maximum normal value; ALT and AST were less than 2.5*maximum normal value; BUN, Cr within 80% of normal range;
7. Patients could understand the circumstances of this study and those who have signed the informed consent form.

Exclusion Criteria:

1. Receive the treatment of other experimental trials in the same period; on the medication of other anticancer drugs at the same time;
2. Patients who have uncontrolled brain metastasis;
3. Suffered from any other malignant tumors in the five years except for complete cure of cervical carcinoma in situ, basal cell cancer;
4. Pregnant or lactating women;
5. Severe infected patients;
6. Patients who have serious cardiovascular disease such as coronary heart disease, unstable cardiac angina and high blood pressure;
7. Patients who have vein thrombus;
8. Patients who have psychiatric illness;
9. Patients who are allergic to E. coli preparation;
10. Researchers believe that those who do not fit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | Assessed up to 24 months
  A duration from date of randomization until the date of first documented progression (as defined by RECIST 1.1) or date of death from any cause, whichever came first. A participant will be censored at the last date they are known not to be progressed.

SECONDARY OUTCOMES:
Objective response rate(ORR) | Assessed up to 24 months
  Objective Response Rate is defined as the proportion of patients with complete response(CR) or partial response(PR) (as defined by RECIST 1.1).
Disease control rate(DCR) | Assessed up to 24 months
  Disease Control Rate is defined as the proportion of patients with complete response(CR), partial response(PR), or stable disease(SD) (as defined by RECIST 1.1).
Overall survival(OS) | Assessed up to 72 months
  Overall Survival is assessed via calculation of the time to death due to any cause. A participant will be censored at the last date they are known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D., Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (37):
- China (37):
  - Bengbu medical college affiliated hospital, Bengbu, Anhui
  - The first affiliated hospital, anhui medical university, Hefei, Anhui
  - The second affiliated hospital, anhui medical university, Hefei, Anhui
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou Medical School, Shantou, Guangdong
  - Guilin medical college affiliated hospital, Guilin, Guangxi
  - The first affiliated hospital of xinxiang medical college, Xinxiang, Henan
  - The Oncology Center of Wuhan Union Hospital, Wuhan, Hubei
  - Zhongnan hospital of Wuhan University, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Yueyang city people's hospital, Yueyang, Hunan
  - The first People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The People 's Liberation Army Eighth Hospital, Nanjing, Jiangsu
  - Affiliate Hospital of Nantong University, Nantong, Jiangsu
  - The first hospital affiliated to suzhou university, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Fourth People's Hospital of Wuxi, Wuxi, Jiangsu
  - Xuzhou medical college affiliated hospital, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - People's hospital SiPingShi center, Siping, Jilin
  - Yanbian university hospital, Yanji, Jilin
  - The tumor hospital of liaoning province, Shenyang, Liaoning
  - Ningxia medical university general hospital, Yinchuan, Ningxia
  - Binzhou medical school affiliated hospital, Binzhou, Shandong
  - Jinan Central Hospital Affiliated of Shandong University, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital ,Sichuan University, Chengdu, Sichuan
  - The second people's hospital of yibin city, Yibin, Sichuan
  - Zhejiang cancer hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No